CLINICAL TRIAL: NCT01196221
Title: Technical Innovation Protocol for Carotid Plaque Imaging by 3.0 Tesla MRI, MRS and Ultrasound: Reproducibility.
Brief Title: Technical Innovation Protocol for MR & US Plaque Imaging: Reproducibility.
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: E.S. stroes, AMC
Other Study IDs: TIP-R
Record Dates: First submitted 2010-09-07; First posted 2010-09-08 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with 30 to 70% carotid artery stenosis

SUMMARY:
The aim of this study is to develop non-invasive MRI, and MRS approaches that will quantify the plaque composition and lipid content of plaques and will have the potential for repeated in vivo measurements. Simultaneously this study aims to develop US plaque imaging as a screening tool to select plaque phenotypes of interest for clinical trials (a large LRNC). For plaque composition imaging by MRI the researchers aim to increase scan resolution and decrease scan time. For quantifying plaque lipid content the researchers aim to develop an MRS protocol. Subsequently, the researchers intend to study the reproducibility of plaque composition and lipid content measurements by MRI, MRS and Ultrasound in subjects that have carotid artery plaques.

ELIGIBILITY:
Inclusion Criteria:

* Patients, with 30 to 70% carotid artery stenosis on ultrasound duplex, who will not go for endarterectomy.

Exclusion Criteria:

* Metal in the body, as a result of e.g. pacemaker or artificial cardiac valves; claustrophobia; surgery performed in the area of measurement (Carotid artery region); Cardiac arrhythmias.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population will consist of patients with carotid artery plaques that cause 30% to 70% lumen stenosis. The degree of stenosis will be assessed by the peak systolic velocity end end diastolic velocity near the stenosis measured by ultrasound duplex.
  The researchers choose to investigate patients with 30% to 70% carotid artery stenosis for the following reasons: 1. Treatment of patients with carotid artery plaques is based on the amount of lumen stenosis. A stenosis of more than 70% is generally treated surgically by endarterectomy. Doing repeated measurements is only possible in patients not treated surgically. 2. Patients with 30% to 70% carotid artery stenosis are, despite their drug treatment, still at high risk for cardiovascular events.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Stroes, MD PhD, Principal Investigator — AIDS Malignancy Consortium
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] Duivenvoorden R, Vanbavel E, de Groot E, Stroes ES, Disselhorst JA, Hutten BA, Lameris JS, Kastelein JJ, Nederveen AJ. Endothelial shear stress: a critical determinant of arterial remodeling and arterial stiffness in humans--a carotid 3.0-T MRI study. Circ Cardiovasc Imaging. 2010 Sep;3(5):578-85. doi: 10.1161/CIRCIMAGING.109.916304. Epub 2010 Jun 24. PMID 20576811